CLINICAL TRIAL: NCT05146401
Title: Associations of Plasma Fatty Acid Patterns During Pregnancy With Gestational Diabetes Mellitus
Brief Title: Associations of Plasma Fatty Acid Patterns With Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Liegang Liu (Other)
Responsible Party: Sponsor-Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: PYL202111
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Gestational Diabetes
Keywords: Fatty acid; Pattern; Gestational diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes mellitus: Gestational diabetes mellitus (GDM) was diagnosed according to the American Diabetes Association criteria, which is based on the "one-step" approach recommended by the International Association of Diabetes and Pregnancy Study Groups. All women underwent a 75g OGTT in the morning after an overnight fast, with plasma glucose measurement fasting and at 1 and 2 hours. The criteria for GDM diagnosis was to have at least one abnormal value: Fasting glucose ≥ 5.1 mmol/L (92 mg/dL), 1 h glucose ≥ 10.0 mmol/L (180 mg/dL), 2 h glucose ≥ 8.5 mmol/L (153 mg/dL).
  Interventions: Other: Plasma fatty acid concentration
- Healthy pregnant women: Pregnant women with fasting glucose < 5.1 mmol/L (92 mg/dL), 1 h glucose < 10.0 mmol/L (180 mg/dL) and 2 h glucose < 8.5 mmol/L (153 mg/dL) were considered as healthy controls. Controls were randomly selected and individually matched to cases by age (± 2 years), gestational age (± 2 weeks) and parity.
  Interventions: Other: Plasma fatty acid concentration

INTERVENTIONS:
Other: Plasma fatty acid concentration — Plasma concentrations of fatty acids were measured by gas chromatography - mass spectrometry (Agilent 7890B gas chromatography coupled with an Agilent 5977A Series mass spectrometry). Individual fatty acids with relative concentrations ≥ 0.05% were used to derive fatty acid patterns through principle components analysis.

SUMMARY:
Background: Limited studies have explored the difference of fatty acid profile between women with and without gestational diabetes mellitus (GDM), and the results were inconsistent. Individual fatty acids tend to be interrelated because of the shared food sources and metabolic pathways. Thus, whether fatty acid patters during pregnancy were related to GDM odds needs further exploration.

Objective: We aim to identify plasma fatty acid patters during pregnancy and their associations with odds of gestational diabetes mellitus (GDM).

Design: A hospital-based case-control study was carried out in urban Wuhan, China from August 2012 to April 2015. Pregnant women who screened for GDM at the outpatient clinics of the Department of Endocrinology, Tongji Hospital were invited to participant in the study. The inclusion criteria were as follows: 1) age ≥ 20 years; 2) gestational age at GDM screening ≥ 24 weeks; 3) singleton pregnancy. We excluded women who met any of the following items: history of diabetes (including but not limited to GDM), cardiovascular disease, cancer or other systemic diseases; pharmacologic treatment or dietary supplement use that might influence glucose or lipids metabolism; accompanied by other pregnancy complications; blood sample hemolysis or insufficiency; incomplete basic information. The diagnosis of GDM can be made if one or more glucose values are above the cut points of 5.1, 10.0 and 8.5 mmol/L at fasting, 1 and 2 h during a 75-gram oral glucose tolerance test (OGTT). Controls were randomly selected and individually matched to cases by age (± 2 years), gestational age (± 2 weeks) and parity. Finally, 217 GDM cases and 217 matched controls were selected in this study. All participants gave written informed consent before enrolling in the study. Fasting blood samples (≥ 8 h overnight fasting) were collected using anticoagulant tubes and centrifuged at 3000 rpm for 5 min. Plasma were separated from blood cells and stored at -80 ℃ for further assay. We measured plasma concentrations of fatty acids by gas chromatography - mass spectrometry, and derived potential fatty acid patterns trough principle components analysis. Conditional logistic regression and restricted cubic spline model were used to evaluate the associations between individual fatty acids or fatty acid patterns and odds of GDM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years;
* Gestational age at GDM screening ≥ 24 weeks;
* Singleton pregnancy;
* With enough plasma collected for fatty acids detection.

Exclusion Criteria:

* History of diabetes (including but not limited to GDM), cardiovascular disease, cancer or other systemic diseases;
* History of receiving pharmacological treatment known to affect glucose metabolism;
* Incomplete basic information.

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the participants enrolled were Chinese women. They gave informed written consent to the study and did not take any medication known to affect glucose tolerance or insulin secretion before participation.
Sampling Method: Probability Sample
Enrollment: 434 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes mellitus | gestation age ≥ 24 weeks
  Glucose intolerance with onset or first diagnosis during pregnancy. The diagnosis of GDM can be made if one or more glucose values are above the cut points of 5.1, 10.0 and 8.5 mmol/L at fasting, 1 and 2 h during a 75-gram oral glucose tolerance test.